CLINICAL TRIAL: NCT04602364
Title: A French Prospective, Observational Cohort Study of Patients With Fabry Disease Treated With Migalastat - the MIGA-FAB Study
Brief Title: French Prospective, Observational Cohort Study of Patients With Fabry Disease Treated With Migalastat
Status: Completed | Type: Observational
Sponsor: Amicus Therapeutics France SAS (Industry)
Responsible Party: Sponsor
Other Study IDs: MIGA-FAB
Record Dates: First submitted 2020-01-22; First posted 2020-10-26 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Miga-Fab patients: Miga-Fab is a French prospective, observational cohort study of patients with Fabry disease treated with migalastat
  Interventions: Other: Noninterventional

INTERVENTIONS:
Other: Noninterventional — Not applicable; Noninterventional study

SUMMARY:
This is a noninterventional cohort study to evaluate the effects of migalastat, on long-term safety, effectiveness, and quality of life (QOL) in patients with Fabry disease.

DETAILED DESCRIPTION:
Occurrence of key indicators of safety and effectiveness will be evaluated, such as cardiac, cerebrovascular and renal events, and overall survival. The study is designed to provide effectiveness and safety data by Q2 2023 which will cover a period up to 5 years after the migalastat launch date.

This will involve a retrospective data collection up to migalastat initiation (for patients already receiving migalastat) and a prospective follow-up from 1 to 3.5 years (depending on the time of enrollment) in migalastat-treated patients with Fabry disease who have a GLA mutation amenable to migalastat.

All visits will be scheduled and conducted according to the clinical site's standard of care. Standard of care is defined as a diagnostic and customary clinical treatment/practice process that a clinician chooses according to their clinical judgement for a Fabry disease patient. There are no study- required visits, tests or clinical assessments.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Fabry disease aged 16 years or older
* eGFRCKD-EPI > 30 mL/min/1.73 m2
* treated with migalastat, or who are starting migalastat upon enrollment
* Patients with Fabry disease and/or parents/guardians (when applicable) who are able to understand and have provided a signed non-opposition form.
* Equipped with a web connection via a computer or tablet

Exclusion Criteria:

* Patients who are participating in a clinical trial of any investigational medicinal product or device at the time of enrollment.
* Patients already included in the present study

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The Miga-Fab is open to participants with Fabry disease treated by migalastat. There is no predetermined sample size.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Safety - SAEs | up to 60 months
  Evaluation of the occurrence ie the number of SAEs
Safety - vital signs | up to 60 months
  Evaluation of resting blood pressure
Effectiveness - Fabry Associated Clinical Events (FACEs) | up to 60 months
  Evaluation of the occurrence of the FACEs ie total number of cardiac, cerebrovascular, and renal events
Effectiveness - survival | From date of inclusion until the date of death from any cause, assessed up to 60 months
  Survival among all patients enrolled, as assessed by recorded patient death from any cause
SF-12 12-Item Short Form Health Survey | up to 60 months
  Evaluation of QOL by the 12-Item Short Form Health Survey (SF-12) ; the higher the score the worse the quality of life is
BPI | up to 60 months
  Brief pain inventory questionnaire ; the higher the score the more intense the pain is
FABPRO-GI | inclusion to last visit
  Fabry Disease Patient-Reported Outcome-Gastro intestinal Signs and Symptoms Questionnaire ; the higher the score the more importante the GI symptoms are
Cardiac echo imagery | up to 60 months
  Echocardiogram (Echo) Left Ventricular Mass Index (LVMI)
Treatment compliance | up to 60 months
  Patient adherence evaluation (% of taken intakes per month) as reported monthly through self-reports of forgotten intakes by the patient

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Lidove, Dr., Principal Investigator — Groupe Hospitalier Diaconnesses Croix Saint Simon
Locations (13):
- France (13):
  - CHU Angers, Angers
  - CHU de Bordeaux, Bordeaux
  - Hôpital Pellegrin, Bordeaux
  - CHU Caen, Caen
  - CHU Lille, Lille
  - Hôpital femme mère enfant, Lyon
  - Hôpital de la Conception | AP-HM, Marseille
  - CHU de Nancy, Nancy
  - CHU Nantes Hôtel Dieu, Nantes
  - Hôpital de la Croix Saint Simon, Paris
  - Hôpital Tenon AP-HP, Paris
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - CHU Toulouse Rangueil, Toulouse

IPD SHARING:
Plan to Share IPD: No